CLINICAL TRIAL: NCT00441519
Title: An Open-Label, Investigator-Blinded, Stratified, Randomized, Parallel Group Study to Compare the Gastroprotective Effects of PA 325 Versus 81 mg Enteric Coated Aspirin
Brief Title: A Parallel Group Study to Compare the Gastroprotective Effects of PA 325 Versus 81 mg Enteric Coated Aspirin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: POZEN (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA325-102
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: Gastroprotective effects; Aspirin
MeSH Terms: interventions — Aspirin; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: aspirin
Drug: omeprazole

SUMMARY:
To compare the gastroprotective effects of a once-daily dose of PA 325 combination tablet

DETAILED DESCRIPTION:
Primary: To compare the gastroprotective effects of a once-daily dose of PA 325 combination tablet combining 325 mg pH sensitive aspirin and 20 mg immediate release omeprazole versus a once-daily dose of 81 mg enteric coated (EC) aspirin utilizing Lanza scores from endoscopy findings in normal healthy volunteers.

Secondary: To evaluate the safety and gastrointestinal tolerability, including ulcerogenic potential, and the effect on gastric pH of PA 325.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or a female who is not pregnant or is not lactating. A female is eligible to enter and participate in this study if she is of:

   * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant); or,
   * Childbearing potential has a negative pregnancy test at screening, and at least one of the following applies or is agreed to by the subject:

     * Complete abstinence from intercourse for at least 14 days prior to first dose of study medication, throughout the study and for 30 days after completion of the study
     * Female sterilization or sterilization of male partner; or,
     * Hormonal contraception by oral route, implant, injectable, vaginal ring; or,
     * Any intrauterine device (IUD) with published data showing that the lowest expected failure rate is less than 1% per year;
     * Double barrier method (2 physical barriers or 1 physical barrier plus spermicide); or
     * Any other method with published data showing that the lowest expected failure rate is less than 1% per year
2. Subject is > 50 years of age inclusive at the time of dosing
3. Subject does not currently smoke and has not smoked for at least 3 months
4. The subject's physical status is within normal limits of age and consistent with observations at screening
5. The subject's Body Mass Index (BMI) is between 20-30 kg/m2
6. Each subject must be able to understand and comply with study procedures required of a subject and is able and willing to provide written informed consent prior to any study procedures being performed

Exclusion Criteria:

1. History of hypersensitivity to omeprazole or to another proton-pump inhibitor
2. History of allergic reaction or intolerance to aspirin or any NSAID and/or a history of NSAID-induced symptoms of asthma, rhinitis, and/or nasal polyps
3. Participation in any study of an investigational treatment in the 4 weeks before Day 1 dosing
4. Presence of uncontrolled acute or chronic medical illness, e.g. GI disorder, hypertension, diabetes, thyroid disorder, depression and/or infection that would endanger a subject if they were to participate in the study
5. GI disorder or surgery leading to impaired drug absorption
6. Evidence of uncontrolled, or unstable cardio- or cerebrovascular disorder, which in the investigator's opinion, would endanger a subject if he or she were to participate in the study
7. Schizophrenia or bipolar disorder
8. Use of any concomitant medication not approved by the study physician during the washout period and during the study conduct
9. Serious blood coagulation disorder, including use of systemic anticoagulants
10. Subjects who donated 50 to 499 mL of blood within 30 days and more than 499 mL within 56 days prior to dosing
11. Subjects who, through completion of the study, would have donated in excess of: 500 mL of blood in 14 days; 1,500 mL of blood in 180 days; 2,500 mL of blood in 1 year
12. Baseline endoscopy showing any gastric or duodenal mucosal abnormality (hemorrhages, ulcers or erosions)
13. Gastric pH > 3 at Day - 1 endoscopy
14. Screening laboratory alanine transaminase (ALT) or aspartate transaminase (AST) value > 2 times the upper limit of normal
15. Estimated creatinine clearance < 30 ml/min at screening
16. Other than noted specifically, any screening laboratory value that is clinically significant in the investigator's opinion and would endanger a subject if he or she were to participate in the study
17. History of hepatitis B or C, a positive test for hepatitis B surface antigen, hepatitis C antibody, a history of HIV infections, or demonstration of HIV antibodies
18. History of malignancy, treated or untreated, within the past 5 years, with the exception of successfully treated basal cell or squamous cell carcinoma of the skin
19. Subjects who have previously been a screen failure in this study
20. Subject has excessive alcohol use (>2 units per day on average; for example 2 bottles of beer, two glasses of wine, 2 ounces of liquor/spirits), or recent history (in the past 3 months) suggestive of alcohol or drug abuse or dependence
21. Subject has ingested grapefruit or grapefruit juice within 10 days of dosing or will ingest grapefruit or grapefruit juice during the duration of the study
22. Positive illicit drug screen

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-02; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the occurrence of gastric and/or duodenal bulb lesions meeting Grade 3 or Grade 4 Lanza (1988) scores for the stomach and duodenal bulb (combined).

SECONDARY OUTCOMES:
Secondary endpoints include the incidence of gastric and/or duodenal ulcers, total number of gastric and/or duodenal erosions, gastric pH and any other GI tolerability issues.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Bryson, Pharm. D., Study Director — POZEN
Locations (2):
- POZEN, Chapel Hill, North Carolina, United States
- MDS Pharma Services, Montreal, Quebec, Canada